CLINICAL TRIAL: NCT02110446
Title: Evaluation of the Efficacy and the Mechanism of Chinese Herbal Formula SS-1 for Sjögren's Syndrome - A Randomized Control Trial
Brief Title: Evaluation of the Efficacy and the Mechanism of Chinese Herbal Formula SS-1 for Sjögren's Syndrome
Acronym: SS-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Chang Gung University (Other); National Science and Technology Council, Taiwan (Other Government); China Medical University, China (Other); China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 102-2481A
Record Dates: First submitted 2014-04-01; First posted 2014-04-10 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Sjögren's Syndrome
Keywords: Sjögren's syndrome; SS-1; Gan-Lu-Yin; Sang-Ju-Yin; Xuefu-Zhuyu-Decoction
MeSH Terms: conditions — Sjogren's Syndrome | interventions — sang ju yin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SS-1 (Experimental): SS-1 is composed of the powder of Gan-Lu-Yin, Sang-Ju-Yin and Xuefu-Zhuyu-Decoction with the ratio of 2:1:1. Patients take 6 gram of experiment medicine three times per day.
  Interventions: Drug: SS-1
- Placebo (Placebo Comparator): The placebo is composed of corn starch, pigment and minimal dose of 1% SS-1. Patients take 6 gram of experiment medicine three times per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SS-1 — The patients will be divided into two groups (A and B) at random and all of them keep the routine treatment in the rheumatology OPD. Group A patients will receive 12 weeks SS-1 treatment first, and then stop the SS-1 for 4 weeks for wash-out phase, and then receive 12weeks placebo treatment. Group B patients receive 12 weeks placebo first, and then stop the placebo treatment for 4 weeks for wash-out phase, and then receive 12weeks SS-1 treatment.
  SS-1 is composed of 3 traditional Chinese herbal formula: Gan-Lu-Yin, Sang-Ju-Yin and Xuefu-Zhuyu-Decoction with the ratio of 2:1:1. The placebo is composed with corn starch, pigment and minimal dose of 1% SS-1. Patients in both groups take 6 gram of SS-1/Placebo three times per day.
  Other Names: Gan-Lu-Yin, Sang-Ju-Yin and Xuefu-Zhuyu-Decoction
  Arms: SS-1
Drug: Placebo — The placebo is composed of corn starch, pigment and minimal dose of 1% SS-1. Patients take 6 gram of experiment medicine three times per day.
  Other Names: 1% SS-1
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of Chinese herbal medicine (SS-1) for the Sjögren's syndrome (SJS) patients.

DETAILED DESCRIPTION:
Investigators take a randomized, double-blinded, placebo-controlled, cross-over design clinical trial to evaluate the effect of Chinese herbal medicine (SS-1) on the regulation of oxidative-related cytokines and the antioxidant capacity for the Sjögren's syndrome (SJS) patients. Through the oxidative stress reduction, the quality of life and clinical manifestation will be improved. Investigators will also use a SJS cell model to elucidate the antioxidant mechanism of SS-1.

The SJS patients in this clinical trial will be screened and be referred from the out-patient department (OPD) of the Rheumatology Department of Chang Gung Memorial Hospital. The patients will be divided into two groups (A and B) at random and all of them keep the routine treatment in the rheumatology OPD. Group A patients will receive 12 weeks SS-1 treatment first and stop the SS-1 for 4 weeks to enter the wash-out phase, and then receive 12 weeks placebo treatment after the wash-out phase. Group B patients receive 12 weeks placebo first and stop the placebo treatment for 4 weeks to enter the wash-out phase, and then receive 12 weeks SS-1 treatment after the wash-out phase. SS-1 is composed of the powder of Gan-Lu-Yin, Sang-Ju-Yin and Xuefu-Zhuyu-Decoction with the ratio of 2:1:1 and the placebo is composed with corn starch, pigment and 1/100 SS-1. Patients in both groups take 6 gram of experiment medicine three times per day. Investigators plan to evaluate the associated parameters at the time just before treatment (V1), after treatment for 12 weeks (V2), at the end of wash-out phase (V3) and when the crossover treatment is completed (V4). Investigators use EULAR Sjogren's syndrome patient reported index, ocular surface disease index and SJS symptom questionnaire for clinical evaluation, and use the SF-36 for quality of life. And investigators use the schirmer's test, salivary scintigraphy, oxidative stress marker and related cytokine for objective observation.

Expected Results:

1. SS-1 may improve the clinical manifestation and quality of life for the patients with Sjögren's syndrome
2. To evaluate the effect of the Chinese medicine on the tongue diagnosis before and after treatment.
3. SS-1 may reduce the oxidative stress (8-OHdG and mtDNA 4977 bp deletion) and elevate the antioxidant capacity (TAC, GSH, mtDNA copy number, SOD, GPX, CAT).
4. SS-1 may have the regulatory effect on cytokine secretion and immune function.
5. SS-1 may have the capacity of reducing the oxidative stress, elevating the antioxidant capacity and regulating the immune response in the model of submaxillary salivary gland cell line with the induction of IFN-γand IFN-α.
6. Identification of the single herb in the SS-1 mixture that regulates oxidative stress and cytokine in the model of submaxillary salivary gland cell line, and set up of the Chinese herbs screen platform for Sjögren's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Primary or Secondary Sjögren's syndrome patient
* Age from 20 to 75 year old, male or female patient
* Fit the criteria of 2002 year American-European classification
* If the subject took Cyclosporine, Cevimeline, Pilocarpine, Rituximab or other biological agent before enter into our study, the subject need to stop these drugs for one month
* If the subject took Gan-Lu-Yin, Sang- Ju-Yin or Xuefu-Zhuyu-Decoction before enter into our study, the subject need to stop these drugs for one month
* Secondary Sjögren's syndrome patient:

  * Stable treatment: Steroid (≦10mg/d) and fixed hydroxychloroquine dose before 3 months enrolled
  * No abnormal change of immunology, liver, kidney, and blood function
  * No major life threatened condition

Exclusion Criteria:

* Alcohol abuse, DM (Glucose PC>200mg/dL) and major life threatened condition
* Pregnancy or breast feeding
* Abnormal liver and kidney function
* Forbid steroid pulse therapy before 3 months enrolled into our study, and forbid the Chinese herbal medicine except SS-1

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Ocular surface disease index (OSDI) | 7 months
  SS-1 may improve the subjective observation of dry eye.
EULAR Sjogren's syndrome patient reported index (ESSPRI) | 7 months
  SS-1 may improve the subjective sensation of dry, pain and fatigue.
SJS symptoms Questionnaire | 7 months
  SS-1 may improve the subjective sensation of dry month.
Schirmer's test | 7 months
  SS-1 may improve the objective observation of dry eye.
Salivary scintigraphy | 7 months
  SS-1 may improve the objective observation of dry month.

SECONDARY OUTCOMES:
Oxidative stress and antioxidant capacity | 7 months
  SS-1 may reduce the oxidative stress and elevate the antioxidant capacity
Quality of life (SF-36) | 7 months
  SS-1 may improve the subjective observation of quality of life.
Regulatory effect on cytokine | 7 months
  SS-1 may have the regulatory effect on cytokine secretion and immune function.

OTHER OUTCOMES:
Adverse effect (AE) and Adverse drug reaction(ADR) | 7 months
  Monitor the Adverse effect (AE) and Adverse drug reaction(ADR) during the SS-1 trial.
Liver, Kidney and Blood function monitor | 7 months
  Monitor the Liver, Kidney and Blood function (RBC, WBC, Hb, PLT, AST, ALT, BUN, Cre) of patient during the SS-1 trial.
Traditional Chinese medicine (TCM) tongue diagnosis | 7 months
  To evaluate the effect of the SS-1 on the TCM tongue diagnosis before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hen-Hong Chang, M.D., Ph.D., Principal Investigator — Chang Gung University
Locations (1):
- Center for Traditional Chinese Medicine, Taoyuan Chang Gung Memorial Hospital, Gueishan Township, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided